CLINICAL TRIAL: NCT06612086
Title: Role of Dapagliflozin in Mangement of Pulmonary Hypertension Patients
Brief Title: Dapagliflozin in Mangement of Pulmonary Hypertension Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, wessam sherif shokry zaki, resident physician of cardiology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dapagliflozin in PH
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Hypertension
Keywords: Dapagliflozin; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Effect of SGLT2 (Dapagliflozin)on prognosis of patient with pulmonary Hypertension and Effect on RV function By speckle tract echocardiography at Assiut University Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- we follow up patient who take Dapagliflozin in patient with pulmonary hypertension (Experimental): we follow up patient who take Dapagliflozin in patient with pulmonary hypertension
  Interventions: Drug: Dapagliflozin (Forxiga)

INTERVENTIONS:
Drug: Dapagliflozin (Forxiga) — we study effect of dapagliflozin on patient with pulmonary hypertension by follow up RV function and prognosis of life of patient

SUMMARY:
Effect of SGLT2 (Dapagliflozin)on prognosis of patient with pulmonary Hypertension and Effect on RV function By speckle tract echocardiography at Assiut University Hospital.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a pathophysiological disorder that may involve multiple clinical conditions and may be associated with a variety of cardiovascular and respiratory diseases. It is clinically diagnosed by a resting mean pulmonary arterial pressure (mPAP) exceeding 20 mmHg . At present, PH's prevalence is approximated at 1 % of the global population and increases to 10 % for individuals over 65 years old, with considerable morbidity and mortality. Sodium-glucose co-transporter 2 inhibitors (SGLT2i) have emerged a metabolic dysfunction and exert cardioprotective effects. DELIVER randomized trials have shown that ( dapagliflozin) can reduce all-cause mortality and hospitalizations due to HF in patients with HF with a mildly reduced or preserved LV function .

The beneficial effects of SGLT2i on the left ventricular systolic and diastolic function, and functional symptom burden have been demonstrated in several studies, but not much is known about the effects of these drugs on the right ventricular (RV) systolic function . The RV is often neglected because of its complex anatomy and the difficulty of obtaining satisfactory imaging "windows" in daily practice . However, the RV has been shown to play an important prognostic role following cardiac surgery and in patients with HF, pulmonary arterial hypertension, or ischemic heart disease . In clinical practice, the assessment of the RV function is usually undertaken by measuring only the longitudinal systolic function, as reflected in the measurement of the tricuspid annular plane systolic excursion (TAPSE) and tricuspid lateral annular systolic velocity (s' wave) derived from Doppler tissue imaging. The fractional area change (FAC), on the other hand, gives us an insight into the radial contraction of the RV [8]. Because these parameters are load- and angle-dependent, advanced echocardiographic methods, such as speckle-tracking echocardiography (STE) measuring the longitudinal strain of the RV free wall (RV FWS) , have recently emerged as more accurate estimates of the RV systolic function . TAPSE and s' wave measure only the longitudinal RV function in the basal region of the RV free wall and were shown to be an independent predictor of cardiac death and major adverse cardiovascular events (MACE) in patients with diverse cardiovascular diseases. Furthermore, the ratio between the TAPSE and systolic pulmonary artery pressure (SPAP) represents the non-invasive measurement of the right ventriculo-arterial coupling and the RV contractile function.

For these reasons, Investigators designed the present study to investigate the effects of SGLT2 espacially dapagliflozin on the RV systolic function after it was added to optimal medical therapy (OMT) on the patient with pulmonary hypertension

ELIGIBILITY:
Inclusion Criteria:

that the patients were diagnosed with pulmonary hypertension By Right heart cath OR suspected By Echocardiograghy according to the ESC guidelines for pulmonary hypertension that they were aged 18 years or older

Exclusion Criteria:

1. symptomatic hypotension (systolic blood pressure < 95 mmHg)
2. impaired renal function (eGFR < 30 mL/min/1.73 m2 calculated according to the CKD-EPI formula) and serum potassium level > 5.2 mmol/L
3. hepatic dysfunction (defined as liver parameters such as ALT, AST, and/or ALP, which are three times above the upper 99-th percentile of the reference range
4. biliary cirrhosis and cholestasis, active malignancies (regardless of the stage and type of malignancy)),
5. the current use of hormone replacement therapy, chemotherapy, or immunotherapy
6. Type 1 diabetes mellitus
7. Acute pulmonary embolism (15)
8. Signficant Primary valvular Heart disease
9. Ischemic heart disease

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Effect of Dapagliflozin on Right ventricle systolic function in patient with pulmonary Hypertension by speckle tract Echocardiography(RV Strain ) | 6 month
  patients with pulmonary hypertension , conventional parameters of RV systolic function, including TAPSE, FAC, s', and RVEF, may be normal despite abnormal RV strain, which is an additional reason for the usage of RV strain in these patients. RV longitudinal strain can identify subclinical RV dysfunction at the early phase of disease and may serve as an important marker of subtle RV systolic dysfunction when conventional parameters, primarily TAPSE, are in the normal range (25, 26).so investigator use RV strain to compare between RV function before and after taking of dapagliflozin

SECONDARY OUTCOMES:
Effect of Dapagliflozin on Quality of life for patient with pulmonary hypertension by Kansas City Cardiomyopathy Questionnaire Score | 6 month
  Quality of the life by Kansas City Cardiomyopathy Questionnaire Score score assess quality of life of patient , investigator used score to compare quality of life before and after taking Dapagliflozin this score are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to100: good to excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Reddy YNV, Carter RE, Sorimachi H, Omar M, Popovic D, Alogna A, Jensen MD, Borlaug BA. Dapagliflozin and Right Ventricular-Pulmonary Vascular Interaction in Heart Failure With Preserved Ejection Fraction: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2024 Sep 1;9(9):843-851. doi: 10.1001/jamacardio.2024.1914. PMID 39046727
- [Background] Li H, Zhang Y, Wang S, Yue Y, Liu Q, Huang S, Peng H, Zhang Y, Zeng W, Wu Z. Dapagliflozin has No Protective Effect on Experimental Pulmonary Arterial Hypertension and Pulmonary Trunk Banding Rat Models. Front Pharmacol. 2021 Nov 1;12:756226. doi: 10.3389/fphar.2021.756226. eCollection 2021. PMID 34790128
- [Background] Kohler S, Zeller C, Iliev H, Kaspers S. Safety and Tolerability of Empagliflozin in Patients with Type 2 Diabetes: Pooled Analysis of Phase I-III Clinical Trials. Adv Ther. 2017 Jul;34(7):1707-1726. doi: 10.1007/s12325-017-0573-0. Epub 2017 Jun 19. PMID 28631216
- [Background] Wang A, Yang K, Wang T, Zhang N, Tang H, Feng X. Effects of sodium-glucose cotransporter 2 inhibitors on risk of venous thromboembolism in patients with type 2 diabetes: A systematic review and meta-analysis. Diabetes Metab Res Rev. 2020 Jan;36(1):e3174. doi: 10.1002/dmrr.3174. Epub 2019 May 27. PMID 31050384
- [Background] Mustapic I, Bakovic D, Susilovic Grabovac Z, Borovac JA. Impact of SGLT2 Inhibitor Therapy on Right Ventricular Function in Patients with Heart Failure and Reduced Ejection Fraction. J Clin Med. 2022 Dec 21;12(1):42. doi: 10.3390/jcm12010042. PMID 36614843
- [Background] Solomon SD, McMurray JJV, Claggett B, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Jhund PS, Belohlavek J, Chiang CE, Borleffs CJW, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer-Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Saraiva JFK, Tereshchenko SN, Thierer J, Vaduganathan M, Vardeny O, Verma S, Pham VN, Wilderang U, Zaozerska N, Bachus E, Lindholm D, Petersson M, Langkilde AM; DELIVER Trial Committees and Investigators. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1089-1098. doi: 10.1056/NEJMoa2206286. Epub 2022 Aug 27. PMID 36027570
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189